CLINICAL TRIAL: NCT02103725
Title: A Phase I, Multi-Centre, Randomised, Vehicle-Controlled, Double-Blinded, Explorative Clinical Trial to Evaluate a Left-Right Design in Adults With Mild to Moderate Atopic Dermatitis Over a Treatment Period of Three Weeks
Brief Title: A Multi-Centre Clinical Trial to Evaluate a Left-Right Design in Adults With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EXP-1092
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pimecrolimus 10 mg/g cream (Experimental): Active drug
  Interventions: Drug: pimecrolimus 10 mg/g cream
- Vehicle cream (Placebo Comparator): Placebo drug
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: pimecrolimus 10 mg/g cream
  Arms: pimecrolimus 10 mg/g cream
Drug: Vehicle cream
  Arms: Vehicle cream

SUMMARY:
The purpose of this study is to validate a left-right design with respect to detecting a difference in efficacy after 3 weeks of treatment between an active treatment and a vehicle in adults with mild to moderate atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female subjects, 18 years or older
* 2. Subject with atopic dermatitis with mild to moderate disease severity
* 3. Two symmetrical and comparable atopic dermatitis treatment areas
* 4. Female volunteers of childbearing potential must either be surgically sterile or agree to use a reliable method of contraception

Exclusion Criteria:

* 1. Any condition in the target areas that in the opinion of the investigator could interfere with clinical assessments, e.g. acne, infection, rash other than atopic dermatitis, sunburn, hyper- or hypopigmentation, scars
* 2. Dark-skinned persons whose skin colour prevents reliable clinical assessments
* 3. Any permanent (or transient within 28 days prior to dosing) disease that may interfere with the subjects safe participation in the trial, with the subjects ability to participate in the trial or with the clinical assessments
* 4. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the treatment effect defined as total sign score on the treated area at end of the 3 weeks treatment period | 3 weeks

SECONDARY OUTCOMES:
Incidence of adverse events during the 3 weeks treatment period | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- bioskin GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en